CLINICAL TRIAL: NCT04465474
Title: Coronavirus Disease 2019 (COVID-19) During Pregnancy: Prevalence of Seroconversion, Effect on Maternal and Perinatal Outcomes and Risk of Vertical Transmission (COVID-MAP)
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Peking University First Hospital (Other); Hospital Universitario de Torrejón (Unknown); Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other); United Christian Hospital (Other); Kwong Wah Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chiu Yee Liona Poon, Prof Poon, Chiu Yee Liona, Chinese University of Hong Kong
Other Study IDs: COVID-MAP
Record Dates: First submitted 2020-07-03; First posted 2020-07-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: pregnancy; vertical transmission; pregnancy loss; ACE2 TMPRSS2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Biological samples Miscarriage: POC, maternal blood
  Stillbirth: Maternal vaginal swab, amniotic fluid, amnion-chorion interface swab, placental tissue, fetal blood, fetal throat swab, maternal blood
  Delivery: Maternal blood before delivery At or after delivery: amniotic fluid, cord blood, placental tissue, amnion-chorion interface swab, neonatal throat swab Breast milk from both breasts for the duration of hospitalization Newborn throat swab at 24 hours of life Newborn stool samples for the duration of hospitalization Infant throat swab and stool sample at 7 days of age Infant blood at 14 days, 6 months & 18 months of age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non Intervention — It's an observational study, no intervention involves.

SUMMARY:
The objectives of this proposal are to: 1) determine the rate of SARS-CoV-2 seroconversion in unselected pregnant women in Hong Kong; 2) determine the rate of SARS-CoV-2 infection in women presenting with miscarriage and stillbirth; 3) follow the pregnancy course and perinatal outcome of confirmed COVID-19-infected pregnant cases; 4) determine the risk and characteristics of vertical transmission; and 5) evaluate the placental barrier, immune response and fetal damage in vertical transmission of SARS-CoV-2. A series of longitudinal and cross-sectional observational studies, and a laboratory-based study will be conducted to fulfil the 5 objectives.

DETAILED DESCRIPTION:
With over 10 million individuals infected worldwide, the coronavirus disease 2019 (COVID-19), caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), is a global public health crisis. It is recognized that pregnant women are at an increased risk of acquiring viral respiratory infection and developing severe pneumonia due to the physiologic changes in their immune and cardiopulmonary systems. Previous studies have attempted to determine maternal and perinatal outcome and potential risk of vertical transmission in pregnant women affected by COVID-19, however, relevant clinical data and biological samples have not been collected in a systematic manner. The research project will engage in collaborative research across obstetricians/maternal-fetal medicine subspecialists, gynecologist, infectious disease specialists, pediatrician, developmental and molecular biologists and bioinformatician between the CUHK, China and Spain. The objectives of this proposal are to: 1) determine the rate of SARS-CoV-2 seroconversion in unselected pregnant women in Hong Kong; 2) determine the rate of SARS-CoV-2 infection in women presenting with miscarriage and stillbirth; 3) follow the pregnancy course and perinatal outcome of confirmed COVID-19-infected pregnant cases; 4) determine the risk and characteristics of vertical transmission; and 5) evaluate the placental barrier, immune response and fetal damage in vertical transmission of SARS-CoV-2. A series of longitudinal and cross-sectional observational studies, and a laboratory-based study will be conducted to fulfil the 5 objectives.

Results generated will inform obstetrics and gynecology, pediatric and infectious disease scientific communities as well as public health specialists and policy makers regarding: (1) the estimated seroconversion rate in women of childbearing age; these results will help (i) improve the approach to care for pregnancy and childbirth during the COVID-19 outbreak; and (ii) formulate preventive measures to be implemented specifically for pregnant women in reducing risk of infection and associated complications to both the women and their unborn child; (2) the impact of COVID-19 on maternal and perinatal outcomes; data from high-quality research will inform practice during the COVID-19 outbreak, guiding healthcare professionals on how to adjust the management approach to infected pregnant women and the exact risks the infection poses to the babies; (3) the risk of vertical transmission at different stages of pregnancy and its sequelae; findings of this study will guide counselling, decision making and clinical management; (4) the identification of cellular site of viral entry and replication in the maternal-fetal interface that would be instrumental in designing therapeutic measures to cease vertical transmission and developing therapeutic treatments.

ELIGIBILITY:
Objective 1: Seroconversion during pregnancy

Inclusion criteria:

* Pregnant women who attended for Down syndrome screening (DSS) at 11-13 weeks
* Had serum sample taken between 1 November 2019 and 1 June 2020 consented for stored serum for future research
* Intended to deliver at the booking hospital.

Objective 2: SARS-CoV-2 and pregnancy loss

Inclusion criteria:

•Pregnant women presenting with first and second trimester miscarriage in Hong Kong and Spain, as well as those with stillbirth during periods of 6 and 12 months, respectively.

Objective 3: Pregnancy course and perinatal outcome

Inclusion criteria:

•Pregnant women affected by COVID-19

Objective 4: Vertical transmission

Inclusion criteria:

•Pregnant women affected by COVID-19

Objective 5: Potential mechanisms for vertical transmission

Inclusion criteria:

•Pregnant women affected by COVID-19

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion during pregnancy - DSS1 | At DSS1 (Around 11-13 weeks gestation)
  Mother
Seroconversion during pregnancy - At delivery | At Delivery
  Mother
Pregnancy loss | At pregnancy loss
  Mother (1st); Mother and abortus/stillborn baby(2nd)
Pregnancy course and perinatal outcome | From date of recruited until the date of delivery
  Mother and Baby
Vertical transmission | At Newborn 0 hours of life, mother immediately after delivery
  Mother and Baby
Vertical transmission | At Newborn 7 days of life
  Mother and Baby
Vertical transmission | At Newborn 14 days of life
  Mother and Baby
Vertical transmission | At Newborn 6 months of life
  Mother and Baby
Vertical transmission | At Newborn 18 months of life
  Mother and Baby
Potential mechanisms for vertical transmission 1) placental barrier, 2) immune response and 3) fetal damage of vertical transmission and mechanism in SARS-CoV-2 infection. | through study completion, up to 2 years
  Mother and Baby

CONTACTS AND LOCATIONS:
Locations (10):
- Peking University First Hospital, Beijing, Beijing Municipality, China
- Hong Kong (8):
  - Kwong Wah Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - United Christian Hospital, Hong Kong
- Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid, Spain

DOCUMENTS (1):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT04465474/Prot_000.pdf